CLINICAL TRIAL: NCT06538701
Title: Effect of Anterolateral Advancement Pharyngoplasty on Retrolingual Collapse in Patients With Multilevel Obstructive Sleep Apnea
Brief Title: Effect of ALA on Retrolingual Collapse in Patients With Multilevel Obstructive OSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Ayman Ahmed Mostafa, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALA in OSA patients
Record Dates: First submitted 2024-07-23; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anterolateral advancement pharyngoplasty (Experimental): Starting with bilateral tonsillectomy, The palatopharyngeal muscle (PPM) raised and advanced to be fixed to the pterygomandibular raphe, The posterior part of the PPM, together with its attached mucosa, was then advanced superolaterally behind the palatoglossus muscle to be hooked up to the levator veli palatini muscle
  Interventions: Procedure: Anterolateral advancement pharyngoplasty

INTERVENTIONS:
Procedure: Anterolateral advancement pharyngoplasty — Starting with bilateral tonsillectomy, The palatopharyngeal muscle (PPM) raised and advanced to be fixed to the pterygomandibular raphe, The posterior part of the PPM, together with its attached mucosa, was then advanced superolaterally behind the palatoglossus muscle to be hooked up to the levator veli palatini muscle

SUMMARY:
To determine the effect of Anterolateral advancement pharyngoplasty on retrolingual collapse in patients with multilevel OSA, and thus if multistage surgery is required.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a condition characterized by repeated episodes of partial or complete airway obstruction during sleep. It is a common health problem affecting a large proportion of the population even among different ethnic groups. At ≥5 events/h apnea-hypopnea index (AHI), the general population prevalence ranged from 9 % to 38 % and was higher in men. The problem increases with advancing age and, in some elderly groups, was as high as 90 % in men and 78 % in women. The prevalence among the adult population ranged from 6 % to 17 % at ≥15 events/h AHI, being as high as 49 % within the advanced ages. The etiology of OSA is multifactorial, consisting of a complex interplay between anatomic, neuromuscular factors and an underlying genetic predisposition toward the disease. Many risk factors have been identified to increase the susceptibility to the disease, including obesity, male sex, ethnicity, and craniofacial structure. The body response to obstructed breathing leads to brain arousal, sympathetic activation, and oxygen desaturation in the blood. This leads to sleep fragmentation, excessive daytime sleepiness and impaired productivity and quality of life (QOL). Obstructive sleep apnea (OSA) has a drastic effect on increasing morbidity and mortality which has been linked to cardiovascular (resistant hypertension, acute myocardial infarction, atrial fibrillation and ventricular tachycardia) and cerebrovascular diseases (stroke, epilepsy and Alzheimer's). Furthermore, OSA has been associated with higher rates of unintentional injury, including motor vehicle collisions and work-related injuries, which add to the public health burden. A polysomnogram (PSG) is an integral component of many sleep evaluations. Attended (Type I) PSGs are the gold standard for diagnosing sleep-related breathing disorders (SRBD), including OSA. The study consists of a simultaneous recording of several physiologic parameters during sleep and wakefulness, including the electroencephalogram (EEG) to identify wake versus sleep and its stages. The main metric for diagnosing OSA in PSG is AHI. According to AHI, the American Academy of Sleep Medicine (AASM) classify the severity of OSA into: Mild with AHI of 5 to <15, moderate with AHI of 15 to 30 and severe with AHI of >30. There are several diagnostic tools which can be useful for the OSA patients' clinical examination, but awake fiberoptic nasopharyngeal endoscopy represents the first level diagnostic technique performed in such patients. The drug-induced sleep endoscopy (DISE) has been introduced to overcome the limits of the awake nasopharyngeal endoscopy. Imaging techniques for diagnosis of OSA include: cephalometric study, fluoroscopy, acoustic reflection, computerized tomography (CT), and magnetic resonance imaging (MRI). Continuous positive airway pressure (CPAP) is the first line treatment option for moderate to severe cases of OSA. CPAP is a highly efficacious therapy for OSA however, poor adherence to therapy can limit the effectiveness of treatment. In OSA patients, obstruction may occur at oropharynx type I, oropharynx and hypopharynx type II, or hypopharynx type III. Most patients have type II obstruction involving both the soft palate and the tongue base. The surgical treatment of OSA patients aimed at widening the diameter of the upper airways by means of resection, advancement and/or suspension, or volumetric reduction of their anatomical structures. Surgical efficacy is linked to the successful identification of the location of the obstruction and its successful correction without causing significant iatrogenic damage, especially if the patient's OSA is not particularly severe. Surgical success is classically defined as a 50% or greater reduction in AHI to less than 20 events per hour. The importance of the lateral pharyngeal wall (LPW) in the pathogenesis of OSA has been demonstrated in a series of articles. In patients with OSA, the LPW is thicker and more collapsible than that of normal subjects when pressured by the airflow. Through progressive increase of positive pressure in a normal subject, enlargement of airway lumen appears mainly in its lateral dimensions, with reduction of thickness of the LPW and with minimal changes in soft palate and tongue. Except when controlling for body mass index (BMI) and neck circumference, LPW narrowing appears to be the sole independent oropharyngeal finding that carries a risk factor for male OSA patients. Uvulopalatopharyngoplasty (UPPP) was first described by akamatsu in 1964, then Fujita introduced it in the USA in 1981. Due to its low success rate and considerable associated complications, the role of this procedure has been questioned, and in the last 2 decades, many modifications of UPPP have been recommended. The recent evolution regarding the techniques of pharyngoplasty has focused on the concept of obtaining expansion and stabilization of the pharyngeal airspace through the treatment of LPW collapse rather than through ablation of redundant pharyngeal soft tissue space. Newer techniques include Lateral pharyngoplasty , Z-palatoplasty, Expansion sphincter pharyngoplasty (ESP) , Relocation pharyngoplasty , Barbed reposition pharyngoplasty (BRP) and, in 2016, Amara et al. described Anterolateral advancement pharyngoplasty (ALA) with no tissue resection nor muscle cutting at all, except for tonsillectomy if not performed before. There are many surgical techniques for retrolingual collapse, they include genioglossus advancement and its different modifications till the more recent one modified genioglossus advancement , radiofrequency tongue base reduction (RFTBR), Tongue base suspension technique and its modifications. Because the airway is a unified system, and the most common cause of retrolingual collapse is glossoptosis caused by negative pressure exerted on the tongue base as a result of palatal and LPW obstruction, relieving obstruction at the palate and LPW will improve obstruction at the tongue base level, eliminating the need for multistage surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 and ≤ 60 years.
* Sex: both genders.
* BMI: less than 32 kg/m2
* Patients with moderate (AHI = 15-30) and severe OSA (AHI > 30) according to the clinical guidelines given by the American Academy of Sleep Medicine
* Friedman tongue position III or IV.
* Documented failure/refusal of attempts of conservative treatment measures (not limited to continuous positive airway pressure).
* The presence of type II obstruction (oropharynx and hypopharynx).
* Class I occlusion.

Exclusion Criteria:

* Age: < 18 or > 60 years old.
* BMI: >32 kg/m2
* Failure to attend postoperative follow-up polysomnography within 12 months of surgery.
* Previous surgery to the base of the tongue or other surgical treatment of OSA.
* Chronic pulmonary disease, or other previous oropharyngeal/laryngeal surgery.
* Class II occlusion with receding mandible.
* Huge lymphoid tissue of the tongue and/or lingual tonsil.
* Symptom not suggestive of OSA and presence of central sleep apnea.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
determine the changes in apnea-hypopnea index (AHI) in multilevel OSA patients with Anterolateral advancement pharyngoplasty | Baseline
  we assess pre- and post-operative polysomnogram to detect if there is changes in AHI (per hour of sleep)
determine the changes in diameter of retrolingual airway in multilevel OSA patients with Anterolateral advancement pharyngoplasty . | Baseline
  we assess pre- and post-operative cephalometry to detect if there is changes in diameter of retrolingual airway (in mm).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed AD Mohammed, proffessor, Study Director — Assiut University

REFERENCES:
- [Background] Cahali MB. Lateral pharyngoplasty: a new treatment for obstructive sleep apnea hypopnea syndrome. Laryngoscope. 2003 Nov;113(11):1961-8. doi: 10.1097/00005537-200311000-00020. PMID 14603056
- [Background] DeRowe A, Gunther E, Fibbi A, Lehtimaki K, Vahatalo K, Maurer J, Ophir D. Tongue-base suspension with a soft tissue-to-bone anchor for obstructive sleep apnea: preliminary clinical results of a new minimally invasive technique. Otolaryngol Head Neck Surg. 2000 Jan;122(1):100-3. doi: 10.1016/S0194-5998(00)70152-5. PMID 10629491
- [Background] Dicus Brookes CC, Boyd SB. Controversies in Obstructive Sleep Apnea Surgery. Sleep Med Clin. 2018 Dec;13(4):559-569. doi: 10.1016/j.jsmc.2018.07.005. PMID 30396449
- [Background] Li HY, Lee LA. Relocation pharyngoplasty for obstructive sleep apnea. Laryngoscope. 2009 Dec;119(12):2472-7. doi: 10.1002/lary.20634. PMID 19688851
- [Background] Powell NB, Riley RW, Guilleminault C. Radiofrequency tongue base reduction in sleep-disordered breathing: A pilot study. Otolaryngol Head Neck Surg. 1999 May;120(5):656-64. doi: 10.1053/hn.1999.v120.a96956. PMID 10229589
- [Background] Riley R, Guilleminault C, Powell N, Derman S. Mandibular osteotomy and hyoid bone advancement for obstructive sleep apnea: a case report. Sleep. 1984;7(1):79-82. doi: 10.1093/sleep/7.1.79. PMID 6718928
- [Background] Vicini C, De Vito A, Benazzo M, Frassineti S, Campanini A, Frasconi P, Mira E. The nose oropharynx hypopharynx and larynx (NOHL) classification: a new system of diagnostic standardized examination for OSAHS patients. Eur Arch Otorhinolaryngol. 2012 Apr;269(4):1297-300. doi: 10.1007/s00405-012-1965-z. Epub 2012 Feb 19. PMID 22350494